CLINICAL TRIAL: NCT03101514
Title: Kanglaite Reduce the Toxicity of Radiotherapy of Head and Neck Cancer Phase II Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201708
Record Dates: First submitted 2017-03-20; First posted 2017-04-05 (Actual); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-02

CONDITIONS: Head and Neck Cancer; Radiotherapy
Keywords: head and neck; tumor; radiotherapy; mucositis; toxicity; Kanglaite injection
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms; Mucositis | interventions — kang-lai-te; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Kanglaite injection + Radiotherapy ± Chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kanglaite group (Experimental): Kanglaite 200ml is injected once a day from Monday to Friday during radiotherapy.
  Interventions: Drug: Kanglaite; Drug: chemotherapy

INTERVENTIONS:
Drug: Kanglaite — Kanglaite injection 200ml is injected intravenous from the first day to the last day of radiotherapy.
  Other Names: Kanglaite injection
Drug: chemotherapy — Cisplatin 80-100mg/m2 was used every 3 weeks during radiotherapy.
  Other Names: Concurrent chemotherapy

SUMMARY:
About 89%-100% patients with head and neck malignant tumors have radiation mucositis during their radiotherapy. Until now, there is no effective method to prevent mucositis. Steroid hormone, pain-relief, anti-inflammatory and other symptom-relief treatments usually are used after the emergence of mucositis. Coixenol triglyceride is an ester extract of Coix Seed. Its trade name is Kanglaite Injection, which has been approved in China and Russia. Kanglaite has anti-tumor effect and reduce treatment toxicity of tumor. Kanglaite could also improve the quality of life of patients and mitigate the condition of the cachexia. In china, two studies evaluating treatment of Kanglaite to nasopharyngeal cancer, found that Kanglaite can reduce radiotherapy mucositis. So far, Kanglaite on the prevention and treatment of radiation mucositis of the head and neck malignant tumor is still lack of strong clinical trial evidence. This is a phase II, single center, one arm study with subject to evaluate the acute radiation mucositis, nutritional status, and quality of life on the course of radiotherapy of head and neck cancer.

DETAILED DESCRIPTION:
3-4 grade radiation mucositis account for 34%-56% in all head and neck patients treated by radiotherapy and >50% in patients treated by radiotherapy concurrent with chemotherapy. 3-4 grade radiation mucositis have obvious symptoms, presenting with fusion ulcers, ulcers bleeding or obvious pain need analgesic drugs. At this time, the patients can not eat or can only intake fluid diet, which led to weight loss, malnutrition, quality of life declined and a series of problems.

Kanglaite has anti-tumor effect and reduce treatment toxicity of tumor. Kanglaite can reduce radiotherapy mucositis of nasopharyngeal cancer had been found initially in Chinese. Kanglaite on the prevention and treatment of radiation mucositis of the head and neck malignant tumor is still lack of strong clinical trial evidence. This is a phase II, single center, one arm study with subject to evaluation the acute radiation mucositis, nutritional status, and quality of life on the course of radiotherapy of head and neck malignant tumors.

Kanglaite 200ml is injected intravenous from the first day to the last day of radiotherapy. Chemotherapy with cisplatin or nedaplatin (both 80-100mg/m2, 21 day per cycle, 1-3 cycles) is used or not concurrent with radiotherapy. There is no order of Kanglaite injection and radiotherapy. Granulocyte colony stimulating factor and antibiotics have no prophylactic use, but can be used after the decline of white blood cells. Mucositis, nutritional status, and quality of life are evaluated before radiotherapy, every week of radiotherapy, 4 weeks after radiotherapy. Mucositis is verified by physical examination. Nutritional status is evaluated by patient-generated subjective global assessment (PG-SGA) scale. Quality of life is evaluated by EORTC QLQ-C30 and QLQ-H&N35 questionnaire.

This is a one arm study, sample size calculation based on the incidence of 3-4 degree mucositis. The incidence of 3-4 degree mucositis is about >50% according to literatures of head and neck squamous cell carcinoma intensity modulated radiation therapy concurrent with chemotherapy. So we assume that Kanglaite can reduce 3-4 degree mucositis from 50% to 30%. The sample size required 44 cases according to the superiority test, bilateral Class I error α = 0.05, class II error β = 0.2. Total 49 cases are need, assuming the off rate of 10%.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old, expected survival period ≥ 12 months
2. Karnofsky score ≥80 points
3. Pathological confirmed head and neck malignant tumors (oral, oropharynx, hypopharynx, throat, nasopharynx, nasal paranasal sinus or other), radical radiotherapy (± chemotherapy) or postoperative radiotherapy (± chemotherapy), radiotherapy dose 60 -70Gy
4. with or without induction chemotherapy (induced chemotherapy ≤ 3 cycles);
5. Meet the following laboratory diagnostic indicators:

   Hemoglobin ≥120g / L, white blood cells 4.0-10.0 × 109 / L, neutrophils 2.0-7.5 × 109 / L, platelets 100-300 × 109 / L; creatinine ≤ normal upper limit (UNL); ALT and AST ≤ 2.5 × UNL, alkaline phosphatase (ALP) ≤ 5 × UNL, total bilirubin (Tbil) ≤ UNL
6. Sign informed consent.

Exclusion Criteria:

1. Distant metastases
2. Allergy to Kanglaite
3. Head and neck had previously received radiation therapy
4. Pregnancy or lactation patients
5. Targeted drug therapy during radiotherapy
6. Radio-chemotherapy uses cytotoxic drugs other than platinum
7. Currently active infections, or combined with rheumatic immune diseases, long-term chronic infection, acute infection, inflammatory state; hematopoietic dysfunction of the blood system diseases; severe cardiopulmonary disease
8. Mental history, can not cooperate with the treatment
9. Researchers believe unsuitable to participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ping Liu, MD, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (1):
- First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No
The investigators have no other clinical trial about cancer of head and neck

REFERENCES:
- [Background] Trotti A, Bellm LA, Epstein JB, Frame D, Fuchs HJ, Gwede CK, Komaroff E, Nalysnyk L, Zilberberg MD. Mucositis incidence, severity and associated outcomes in patients with head and neck cancer receiving radiotherapy with or without chemotherapy: a systematic literature review. Radiother Oncol. 2003 Mar;66(3):253-62. doi: 10.1016/s0167-8140(02)00404-8. PMID 12742264
- [Background] Redding SW. Cancer therapy-related oral mucositis. J Dent Educ. 2005 Aug;69(8):919-29. PMID 16081575
- [Background] Silverman S Jr. Diagnosis and management of oral mucositis. J Support Oncol. 2007 Feb;5(2 Suppl 1):13-21. PMID 17366929
- [Background] Harris DJ. Cancer treatment-induced mucositis pain: strategies for assessment and management. Ther Clin Risk Manag. 2006 Sep;2(3):251-8. doi: 10.2147/tcrm.2006.2.3.251. PMID 18360600
- [Background] Rodriguez-Caballero A, Torres-Lagares D, Robles-Garcia M, Pachon-Ibanez J, Gonzalez-Padilla D, Gutierrez-Perez JL. Cancer treatment-induced oral mucositis: a critical review. Int J Oral Maxillofac Surg. 2012 Feb;41(2):225-38. doi: 10.1016/j.ijom.2011.10.011. Epub 2011 Nov 8. PMID 22071451
- [Background] Walsh L, Gillham C, Dunne M, Fraser I, Hollywood D, Armstrong J, Thirion P. Toxicity of cetuximab versus cisplatin concurrent with radiotherapy in locally advanced head and neck squamous cell cancer (LAHNSCC). Radiother Oncol. 2011 Jan;98(1):38-41. doi: 10.1016/j.radonc.2010.11.009. Epub 2010 Dec 13. PMID 21159400
- [Background] Chen Y, Liu MZ, Liang SB, Zong JF, Mao YP, Tang LL, Guo Y, Lin AH, Zeng XF, Ma J. Preliminary results of a prospective randomized trial comparing concurrent chemoradiotherapy plus adjuvant chemotherapy with radiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma in endemic regions of china. Int J Radiat Oncol Biol Phys. 2008 Aug 1;71(5):1356-64. doi: 10.1016/j.ijrobp.2007.12.028. Epub 2008 May 9. PMID 18472356
- See also: Jing JL, Li XL, Nan YQ. Advances in the study of the effect of Kanglaite injection on tumor therapy. Chinese Remedies & Clinics, 2013;13(11):1447-1448 (in Chinese). — http://www.cnki.net/KCMS/detail/detail.aspx?QueryID=1&CurRec=1&filename=YWLC201311028&dbname=CJFD2013&dbcode=CJFQ&pr=&urlid=&yx=&uid=WEEvREcwSlJHSldRa1FhdkJkcGkzcVBMVDlLcXRDRGlQd3hhNzRBZkFjbz0=$9A4hF_YAuvQ5obgVAqNKPCYcEjKensW4IQMovwHtwkF4VYPoHbKxJw!!&v=MTgzNDJDVVJMMmZaT1J2Rml6Z1ViN0FQRHJIYmJHNEg5TE5ybzlIYklSOGVYMUx1eFlTN0RoMVQzcVRyV00xRnI=
- See also: Guo Y, Li DP. Protective effects of Kanglaite injection on hematopoiesis and liver and kidney damage caused by three anticancer drugs. Chinese journal of modern applied phaemacy.1998;15(6):61-62(in Chinese). — http://www.cnki.net/KCMS/detail/detail.aspx?QueryID=6&CurRec=1&filename=XDYD199806032&dbname=CJFD9899&dbcode=CJFQ&pr=&urlid=&yx=&uid=WEEvREcwSlJHSldRa1FhdkJkcGkzcVBMVDlLcXRDRGlQd3hhNzRBZkFjbz0=$9A4hF_YAuvQ5obgVAqNKPCYcEjKensW4IQMovwHtwkF4VYPoHbKxJw!!&v=MjczNDlPUnZGaXpnVkx6QVBTblNhckt4RjluTXFZOUdab1I4ZVgxTHV4WVM3RGgxVDNxVHJXTTFGckNVUkwyZlo=
- See also: Wang WD, Sun SP, Wang XD. Influence of KLT on Radiotherapy Effect of Patients with Advanced Nasopharyngeal Carcinoma. China Journal of Cancer Prevention and Treatment,2003:10(6): 635-637(in Chinese). — http://www.cnki.net/KCMS/detail/detail.aspx?QueryID=0&CurRec=1&filename=QLZL200306029&dbname=CJFD2003&dbcode=CJFQ&pr=&urlid=&yx=&uid=WEEvREcwSlJHSldRa1FhdkJkcGkzcVBMVDlLcXRDRGlQd3hhNzRBZkFjbz0=$9A4hF_YAuvQ5obgVAqNKPCYcEjKensW4IQMovwHtwkF4VYPoHbKxJw!!&v=MDkyNDc0SHRMTXFZOUhiWVI4ZVgxTHV4WVM3RGgxVDNxVHJXTTFGckNVUkwyZlpPUnZGaS9rVnIvSk5DSFJZckc=
- See also: Ren ZP, et al. The therapeutic effects of the combined therapy with kanglaite injection and radiotherapy on nasopharyngea carcinoma among aged cases. Chinese Journal of Otorhinolaryngology of Integrated Traditional and Western Medici 2005;13(6) — http://www.cnki.net/KCMS/detail/detail.aspx?QueryID=0&CurRec=1&filename=XYJH200506008&dbname=CJFD2005&dbcode=CJFQ&pr=&urlid=&yx=&uid=WEEvREcwSlJHSldRa1FhdkJkcGkzcVBMVDlLcXRDRGlQd3hhNzRBZkFjbz0=$9A4hF_YAuvQ5obgVAqNKPCYcEjKensW4IQMovwHtwkF4VYPoHbKxJw!!&v=MDM5ODBlWDFMdXhZUzdEaDFUM3FUcldNMUZyQ1VSTDJmWk9SdkZpL2xWYnZBUFRUQlpyRzRIdFRNcVk5RmJJUjg=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited patients with head and neck cancer receiving radiotherapy in the First Affiliated Hospital of Harbin Medical University between January 2017 and October 2019.
Pre-assignment Details: Sixty-two patients were assessed for eligibility. Three patients did not meet the inclusion criteria, and six patients declined to participate.
Groups:
- Kanglaite Group: All patients received 20 g Kanglaite (200 mL) daily, administered as an intravenous injection for 5 days a week, concurrently with radiotherapy. Kanglaite injection was used before or after radiotherapy. There is no time interval requirement between Kanglaite and radiotherapy.
Period: Overall Study
Arm/Group | Kanglaite Group
Started | 53
Completed | 46
Not Completed | 7
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 2
Not completed — patient's information was incomplete | 1

BASELINE CHARACTERISTICS:
Groups:
- Kanglaite Group: Kanglaite injection was used during radiotherapy
Arm/Group | Kanglaite Group
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 46
Nutritional status [Count of Participants; unit: Participants] — Nutritional status was scored using Patient-Generated Subjective Global Assessment (PG-SGA) questionnaire.A score of 0-1 indicated good nourishment, a score of 2-8 indicated suspected or moderate malnutrition, and a score ≥ 9 indicated risk of severe malnutrition.
  Participants
    Severe malnutrition | 9
    Suspected or moderate malnutrition | 31
    Good nourishment | 6
Quality of life specific to head and neck cancers [Mean (Standard Deviation); unit: units on a scale] — Quality of life specific to head and neck cancers was assessed by EORTC-QLQ-H&N35 questionnaires. Each item of the QLQ-H&N35 was scored from 0 to 100. Higher scores indicated a worsening quality of life.
  units on a scale
    pain | 19.22 (25.15)
    swallowing | 16.62 (24.08)
    sensory problems | 9.25 (22.34)
    speech problems | 25.67 (29.28)
    social eating problems | 14.43 (25.95)
    social contact problems | 9.48 (19.70)
    less sexuality | 17.55 (30.89)
    teeth | 24.44 (32.09)
    mouth opening problem | 11.58 (24.77)
    dry mouth | 22.22 (26.59)
    sticky saliva | 30.36 (31.64)
    coughing | 22.22 (28.42)
    feeling ill | 22.22 (27.52)
Overall quality of life (QOL) [Mean (Standard Deviation); unit: units on a scale] — Overall quality of life was assessed by EORTC-QLQ-C30 questionnaires.Each item of the QLQ-C30 was scored from 0 to 100. Higher scores for function on the QLQ-C30 (global QOL, physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning) indicated a better QOL, whereas higher scores for the symptoms on the QLQ-C30 (fatigue, nausea and vomiting, pain, dyspnoea,insomnia, appetite loss,constipation, diarrhoea) indicated a worsening QOL
  units on a scale
    global QOL | 73.18 (25.39)
    physical functioning | 89.99 (12.05)
    role functioning | 82.6 (24.33)
    emotional functioning | 84.48 (18.36)
    cognitive functioning | 81.46 (25.92)
    social functioning | 71.1 (30.02)
    fatigue | 21.40 (19.34)
    nausea and vomiting | 4.07 (12.38)
    pain | 16.3 (19.29)
    dyspnoea | 12.59 (22.79)
    insomnia | 14.07 (27.05)
    appetite loss | 14.81 (25.18)
    constipation | 10.36 (21.10)
    diarrhoea | 8.88 (16.51)

OUTCOME MEASURES:

1. Primary Outcome: the Incidence Rate of Severe Radiation Mucositis
Description: The grade of radiation mucositis was assessed by CTCAE v4. The highest grade be recorded. The grade 1 was the best and grade 4 was the worst.
Time Frame: From date of randomization until the end radiotherapy, up to 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Kanglaite Group
Number analyzed (Participants) | 46
Participants
  Grade 1 mucositis | 3
  Grade 2 mucositis | 38
  Grade 3 mucositis | 5
  Grade 4 mucositis | 0

2. Secondary Outcome: the Incidence Rate of Non-Hematologic Toxicity Side Events
Description: The non-hematologic toxicity side events were assessed by CTCAE v4. The highest grade be recorded. The grade 1 was the best and grade 4 was the worst.
Time Frame: From date of randomization until the end radiotherapy, up to 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Kanglaite Group
Number analyzed (Participants) | 46
Participants
  grade 1 superficial phlebitis | 1
  grade 1 rash | 1
  radiotherapy dose reduction | 1
  irradiation field modification | 0
  radiotherapy interruption | 4

3. Secondary Outcome: the Incidence Rate of Hematologic Toxicity Side Events
Description: The grade of hematologic toxicity side events were assessed by CTCAE v4. The highest grade be recorded. The grade 1 was the best and grade 4 was the worst.
Time Frame: From date of randomization until the end radiotherapy, up to 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Kanglaite Group
Number analyzed (Participants) | 46
Participants
  Neutropenia: grade 0 | 30
  Neutropenia: grade 1-2 | 13
  Neutropenia: grade 3-4 | 3
  Anemia: grade 0 | 28
  Anemia: grade 1-2 | 18
  Anemia: grade 3-4 | 0
  Thrombocytopenia: grade 0 | 40
  Thrombocytopenia: grade 1-2 | 6
  Thrombocytopenia: grade 3-4 | 0
  Pre-albumin decrease: grade 0 | 37
  Pre-albumin decrease: grade 1-2 | 9
  Pre-albumin decrease: grade 3-4 | 0
  Albumin decreasing: grade 0 | 44
  Albumin decreasing: grade 1-2 | 2
  Albumin decreasing: grade 3-4 | 0
  alanine transaminase increasing: grade 0 | 41
  alanine transaminase increasing: grade 1-2 | 5
  alanine transaminase increasing: grade 3-4 | 0
  aspartate transaminase increasing: grade 0 | 43
  aspartate transaminase increasing: grade 1-2 | 3
  aspartate transaminase increasing: grade 3-4 | 0
  alkaline phosphatase increasing: grade 0 | 45
  alkaline phosphatase increasing: grade 1-2 | 1
  alkaline phosphatase increasing: grade 3-4 | 0
  total bilirubin increasing: grade 0 | 43
  total bilirubin increasing: grade 1-2 | 3
  total bilirubin increasing: grade 3-4 | 0
  creatinine increasing: grade 0 | 44
  creatinine increasing: grade 1-2 | 2
  creatinine increasing: grade 3-4 | 0
  blood urea nitrogen increasing: grade 0 | 45
  blood urea nitrogen increasing: grade 1-2 | 1
  blood urea nitrogen increasing: grade 3-4 | 0

4. Secondary Outcome: the Nutritional Status
Description: The nutritional status was assessed by PG-SGA questionnaire.PG-SGA scores were recorded weekly during radiotherapy. A score of 0-1 indicated good nourishment, 2-8 suspected or moderate malnutrition, ≥ 9 risk of severe malnutrition.
Time Frame: From date of randomization until the end radiotherapy, up to 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Kanglaite Group
Number analyzed (Participants) | 46
Participants
  Score 0-1 | 2
  Score 2-8 | 13
  Score ≧9 | 31

5. Secondary Outcome: the Overall Quality of Life (QOL)
Description: The overall quality of life was assessed by EORTC QLQ-C30 questionnaire. QLQ-C30 scores were valued weekly during radiotherapy and post radiotherapy.The worst score of patients was recorded. The QLQ-C30 was scored from 0 to 100. Higher scores for function indicated a better QOL whereas the symptoms indicated a worsening QOL.
Time Frame: From date of randomization until the end radiotherapy, up to 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Kanglaite Group
Number analyzed (Participants) | 46
units on a scale
  global quality of life during radiotherapy | 56.52 (29.80)
  physical functioning during radiotherapy | 77.19 (21.66)
  rolel functioning during radiotherapy | 70.28 (27.42)
  emotional functioning during radiotherapy | 77.35 (22.07)
  cognitive functioning during radiotherapy | 74.99 (23.23)
  social functioning during radiotherapy | 62.68 (31.26)
  fatigue during radiotherapy | 32.32 (21.91)
  nausea and vomiting during radiotherapy | 22.07 (24.09)
  pain during radiotherapy | 34.05 (26.73)
  dyspnoea during radiotherapy | 21.01 (28.42)
  insomnia during radiotherapy | 31.15 (31.74)
  appetite loss during radiotherapy | 43.47 (32.10)
  costipation during radiotherapy | 26.08 (28.90)
  diarrhoea during radiotherapy | 12.31 (19.06)
  global quality of life post radiotherapy | 64.72 (24.93)
  physical functioning post radiotherapy | 81.09 (22.00)
  role functioning post radiotherapy | 75.58 (25.02)
  emotional functioning post radiotherapy | 97.4 (10.47)
  cognitive functioning post radiotherapy | 83.72 (20.72)
  social functioning post radiotherapy | 72.09 (27.39)
  fatigue post radiotherapy | 28.16 (23.30)
  nausea and vomiting post radiotherapy | 11.26 (19.08)
  pain post radiotherapy | 21.70 (23.43)
  dyspnoea post radiotherapy | 19.12 (31.82)
  insomnia post radiotherapy | 21.70 (30.67)
  appetite post radiotherapy | 39.53 (30.21)
  constipation post radiotherapy | 16.27 (23.42)
  diarrhoea post radiotherapy | 4.65 (11.68)

6. Secondary Outcome: Quality of Life Specific to Head and Neck Cancers
Description: Quality of life specific to head and neck cancers was assessed by EORTC QLQ-H&N35 questionnaire. QLQ-H&N35 scores were valued weekly during radiotherapy and post radiotherapy. The highest score of patients was recorded. The QLQ-H&N35 was scored from 0 to 100. Higher scores indicated a worsening QOL.
Time Frame: From date of randomization until the end radiotherapy, up to 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Kanglaite Group
Number analyzed (Participants) | 46
units on a scale
  pain during radiotherapy | 41.83 (23.72)
  swallowing during radiotherapy | 42.03 (27.05)
  sensory problems during radiotherapy | 35.5 (26.89)
  speech problems during radiotherapy | 43.59 (36.51)
  social eating problems during radiotherapy | 40.57 (30.51)
  social contact problems during radiotherapy | 21.08 (25.52)
  less sexuality during radiotherapy | 41.86 (40.67)
  teeth during radiotherapy | 28.98 (34.14)
  mouth opening problems during radiotherapy | 27.53 (28.37)
  dry mouth during radiotherapy | 60.14 (29.49)
  sticky saliva during radiotherapy | 66.66 (26.29)
  coughing during radiotherapy | 42.75 (33.45)
  feeling ill during radiotherapy | 47.40 (27.05)
  pain post radiotherapy | 33.72 (26.11)
  swallowing post radiotherapy | 36.04 (23.40)
  sensory problems post radiotherapy | 36.04 (29.30)
  speech problems post radiotherapy | 38.49 (35.41)
  social eating problems post radiotherapy | 28.09 (24.60)
  social contact problems post radiotherapy | 11.99 (17.03)
  less sexuality post radiotherapy | 37.96 (38.34)
  teeth post radiotherapy | 23.25 (29.57)
  mouth opening problems post radiotherapy | 12.40 (17.85)
  dry mouth post radiotherapy | 53.48 (34.22)
  sticky saliva post radiotherapy | 56.58 (35.28)
  coughing post radiotherapy | 37.2 (33.49)
  feeling ill post radiotherapy | 37.20 (29.28)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Kanglaite Group
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 7/46
Other Adverse Events (participants affected / at risk) | 34/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kanglaite Group (N=46)
mucositis (Skin and subcutaneous tissue disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Kanglaite Group (N=46)
anemia (Blood and lymphatic system disorders) | 18
Neutropenia (Blood and lymphatic system disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Pre-albumin (General disorders) | 9
Alanine aminotransferase (Hepatobiliary disorders) | 5
Glutamic oxaloacetic transaminase (Hepatobiliary disorders) | 3
Total bilirubin (Hepatobiliary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT03101514/Prot_SAP_000.pdf